CLINICAL TRIAL: NCT02800486
Title: Phase II Trial of Super Selective Intra-arterial Repeated Infusion of Cetuximab (Erbitux) With Reirradiation for Treatment of Relapsed/Refractory Glioblastoma Multiforme, Anaplastic Astrocytoma, and Anaplastic Oligoastrocytoma
Brief Title: Super Selective Intra-arterial Repeated Infusion of Cetuximab (Erbitux) With Reirradiation for Treatment of Relapsed/Refractory GBM, AA, and AOA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS16-0181
Record Dates: First submitted 2016-05-27; First posted 2016-06-15 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma; Anaplastic Astrocytoma; Anaplastic Oligoastrocytoma; Glioma; Brain Neoplasm; Brain Cancer; Brain Tumor; Brain Tumor, Recurrent; Brain Neoplasm, Malignant
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra-arterial Cetuximab with Re-Irradiation (Experimental): Mannitol 20% 12.5ml over two minutes for blood brain barrier (BBB) disruption followed by Cetuximab administered intra-arterially for three doses at a dose of 250 mg/m2 combined with hypofractionated re-irradiation
  Interventions: Drug: Intra-arterial Cetuximab; Drug: Intra-arterial Mannitol; Radiation: Hypofractionated re-irradiation

INTERVENTIONS:
Drug: Intra-arterial Cetuximab
Drug: Intra-arterial Mannitol
Radiation: Hypofractionated re-irradiation

SUMMARY:
Primary brain tumors are typically treated by surgery, radiation therapy and chemotherapy, either individually or in combination. Present therapies are inadequate, as evidenced by the low 5-year survival rate for brain cancer patients, with median survival at approximately 12 months. Glioma is the most common form of primary brain cancer, afflicting approximately 7,000 patients in the United States each year. These highly malignant cancers remain a significant unmet clinical need in oncology. GBM often has a high expression of EFGR (Epidermal Growth Factor Receptor), which is associated with poor prognosis. Several methods of inhibiting this receptor have been tested, including monoclonal antibodies, vaccines, and tyrosine kinase inhibitors. The investigators hypothesize that in patients with recurring GBM, intracranial superselective intra-arterial infusion of Cetuximab (CTX), at a dose of 250mg/m2 in conjunction with hypofractionated radiation, will be safe and efficacious and prevent tumor progression in patients with recurrent, residual GBM.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of ≥18 years of age
* Patients with a documented histologic diagnosis of relapsed or refractory glioblastoma multiforme (GBM), anaplastic astrocytoma (AA) or anaplastic oligoastrocytoma (AOA)
* Patients with pathology confirmed histologic EGFR overexpression
* Patients must have at least one confirmed and evaluable tumor site.∗

  *A confirmed tumor site is one in which is biopsy-proven
* Patients must have a Karnofsky performance status ≥60% and an expected survival of ≥ three months.
* No chemotherapy for two weeks prior to treatment under this research protocol and no external beam radiation for eight weeks prior to treatment under this research protocol
* Patients must have adequate hematologic reserve with WBC≥3000/mm3, absolute neutrophils ≥1500/mm3 and platelets ≥100,000/ mm3. Patients who are on Coumadin must have a platelet count of ≥150,000/ mm3
* Pre-enrollment chemistry parameters must show: bilirubin<1.5X the institutional upper limit of normal (IUNL); AST or ALT<2.5X IUNL and creatinine<1.5X IUNL
* Pre-enrollment coagulation parameters (PT and PTT) must be ≤1.5X the IUNL
* Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study
* Patients must be able to understand and give written informed consent. Informed consent must be obtained at the time of patient screening

Exclusion Criteria:

* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men will be informed of the potential unknown risk of conception while participating in this research trial and will be advised that they must use effective contraception during and for a period of three months after the treatment period
* Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring
* Patients with radiological evidence of leptomeningeal disease
* Patients with history of allergic reaction to CTX
* Patients who completed chemo/RT less than 6 months prior to enrollment
* Patients who have not failed standard Stupp protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 6 months
  The 6-month PFS will be estimated by calculating the proportion of patients who are alive at 6 months from treatment commencement and are progression-free.
Overall Survival (OS) | 2 years
  OS will be calculated as the time from treatment initiation to the date of death.

SECONDARY OUTCOMES:
Composite overall response rate (CORR) through the Response Evaluation Criteria In Solid Tumors (RECIST) | 6 months
  Subjects will be classified according to the RECIST criteria, which is a composite of MRI changes, clinical response and changes in steroid use.
Toxicities graded according to the NCI Common Toxicity Criteria (CTCAE) version 4.03 | 6 months
  Toxicities will be tabulated and graded according to the NCI Common Toxicity Criteria (CTCAE) version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Northwell Health
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No